CLINICAL TRIAL: NCT03372577
Title: Mindfulness-based Sex Therapy on Patients With Takotsubo Cardiomyopathy Among Iranian Women
Brief Title: Mindfulness-based Sex Therapy on Patients With Takotsubo Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Director of Social Determinants of Health Research Center (SDH), Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.QUMS.REC.1396.188
Record Dates: First submitted 2017-12-09; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Takotsubo Cardiomyopathy; Sexual Dysfunction
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Sexual Dysfunction, Physiological | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patient and partner (Experimental)
  Interventions: Behavioral: Mindfulness-Based Sex Therapy
- patient ,partner and cardiac rehabilitation team (Experimental)
  Interventions: Behavioral: Mindfulness-Based Sex Therapy
- Treatment as usual (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-Based Sex Therapy — It is based on an integration of psychoeducation, sex therapy, and mindfulness-based skills. the intervention will be delivered by a group of facilitators on a group based weekly.
  Arms: patient ,partner and cardiac rehabilitation team; patient and partner
Other: Treatment as usual — Routine discharge counseling
  Arms: Treatment as usual

SUMMARY:
Takotsubo cardiomyopathy (TC) is a type of non-ischemic cardiomyopathy in which there is a sudden temporary weakening of the myocardium. . In a recent study, women report more sexual dysfunction than men after 1 year after TC. Despite that a number of studies have assessed female sexual dysfunction (FSD) for TC , there is no information regarding prevalence and associated factors on FSD in women with TC. However, in a recent study on Iranian female patients with TC, more than 77% of these patients suffered from FSD. This study is aimed to assess the effectiveness of a Mindfulness-based Sex Therapy on Patients With TC.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years old at least
* confirmed diagnosis of TC by a cardiologist according Mayo Clinic diagnostic criteria; an acute left ventricular apical ballooning of unknown cause
* willingness to partaking for the duration of the trial
* a basic fluency in Persian
* living with a partner/spouse

Exclusion Criteria:

* cognitive disability
* having acute myocardial infarction
* cerebrovascular disease
* pheochromocytoma and viral or idiopathic myocarditis
* , participating in another RCT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Sexual functioning | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Sexual functioning is assessed using self-reported measure , female Sexual Function Index (FSFI)
Sexual Distress | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Female Sexual Distress Scale;The FSDS-R is a self-reported questionnaire consisting of 13 items assessing different aspects of sexual activity-related distress in women
Intimacy | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Personal Assessment of Intimacy in Relationships (PAIR) will use to assess relationship satisfaction. The PAIR is a self-reported measure with 36 items which cover five subscales

SECONDARY OUTCOMES:
Mindfulness | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Sexual Five-Facet Mindfulness Questionnaire (FFMQ-S) is used to assess mindfulness in the context of sexual encounters
Marital satisfaction | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  The Maudsley Marital Questionnaire (MMQ) is a 20-item instrument measuring marital satisfaction.
Psychological distress | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Hospital Anxiety and Depression Scale (HADS) is a brief self-administrated tool to assess psychological distress in patients as well as general populations
Rumination | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Rumination is measured using Ruminative Thought Style Questionnaire (RTS). The RTS contains 20 items describing positive, negative and neutral facets of global rumination
Emotion regulation | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Persons' emotions in response to stressful life events is measured using he Cognitive Emotion Regulation Questionnaire short version (CERQ-short).
quality of life | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  HRQoL is measured using Short Form health survey (SF-12).
Social Support | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Social support will be assessed by the ENRICHD Social Support Inventory (ESSI ).
Sense of Coherence | changes from baseline, 1 Months ,6 months, 12 months and 18 months
  Sense of coherence will be measured using the Antonovsky's 13-item sense of coherence scale (SOC-13).

CONTACTS AND LOCATIONS:
Locations (1):
- Booali Sina Hospital, Qazvin, Iran

IPD SHARING:
Plan to Share IPD: Undecided